CLINICAL TRIAL: NCT01850797
Title: Registry of Acute Stroke Under New Oral Anticoagulants -Pilot (RASUNOA-Pilot)
Acronym: RASUNOA
Status: Completed | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Prof. Roland Veltkamp, Senior Physician, Department of Neurology, University Hospital Heidelberg, University Hospital Heidelberg
Other Study IDs: S-556/2011
Record Dates: First submitted 2013-05-07; First posted 2013-05-09 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Ischemic Stroke; Intracranial Hemorrhage
Keywords: oral anticoagulants; ischemic stroke; blood thinner; intracranial hemorrhage
MeSH Terms: conditions — Ischemic Stroke; Intracranial Hemorrhages

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NOAC: Patients receiving NOAC and suffering from ischemic stroke or intracranial bleeding.

SUMMARY:
The registry of acute stroke under new oral anticoagulants (RASUNOA) is a German multicenter, prospective, observational registry performed at about 50 study centers covering about 50.000 acute ischemic strokes and 6000 acute intracranial hemorrhages per year. Study enrollment will be consecutive. The RASUNOA registry study center is the University Medical Center of the Principal Investigator (Heidelberg, Germany). The registry will focus on treatment decisions and concepts in patients being under treatment with a new oral anticoagulant and suffering from acute ischemic or hemorrhagic stroke.

DETAILED DESCRIPTION:
The main purpose of the study is to collect information from a large, prospectively enrolling multicentre stroke database regarding the optimal management of ischemic and hemorrhagic stroke during anticoagulation with nOAC. Specifically, we aim to obtain critical information regarding the epidemiology, natural history, laboratory and neuroradiological aspects, clinical consequences, and the effects of treatment (i.e. thrombolysis/interventional recanalisation in ischemic stroke and hemostatic therapy in ICH, respectively) in stroke during nOAC. The Registry is not limited to a specific new OAC but intends to examine stroke during use of any of the approved nOAC. The study is not designed to perform comparisons among the different nOAC.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 years
* informed consent
* acute stroke or intracranial bleeding
* therapy with a new oral anticoagulant (Dabigatran®, Rivaroxaban®, Apixaban®, Edoxaban®)

Exclusion Criteria:

* missing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients suffering from acute ischemic stroke or intracranial hemorrhage while being anti coagulated. Only patients taking new oral anticoagulants will be included.
Sampling Method: Non-Probability Sample
Enrollment: 353 (Actual)
Dates: Start 2012-01; Primary Completion 2015-03 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Rate of hematoma expansion (ICH) | 48h after ICH
  Rate of hematoma enlargement in patients with ICH between initial imaging and follow-up imaging (CT)
Symptomatic intracerebral haemorrhage after thrombolysis | 24 h
  In patients with ischemic stroke while under treatment with any of the new OAC who receive thrombolysis we will measure any hemorrhagic transformation on routine follow-up CT imaging (usually within 24h after thrombolysis)

CONTACTS AND LOCATIONS:
Overall Officials: Roland Veltkamp, Prof., Principal Investigator — University Hospital Heidelberg
Locations (1):
- University Hospital Heidelberg, Heidelberg, Germany

REFERENCES:
- [Derived] Purrucker JC, Haas K, Rizos T, Khan S, Poli S, Kraft P, Kleinschnitz C, Dziewas R, Binder A, Palm F, Jander S, Soda H, Heuschmann PU, Veltkamp R; RASUNOA Investigators (Registry of Acute Stroke Under New Oral Anticoagulants). Coagulation Testing in Acute Ischemic Stroke Patients Taking Non-Vitamin K Antagonist Oral Anticoagulants. Stroke. 2017 Jan;48(1):152-158. doi: 10.1161/STROKEAHA.116.014963. Epub 2016 Nov 29. PMID 27899756
- [Derived] Purrucker JC, Wolf M, Haas K, Rizos T, Khan S, Dziewas R, Kleinschnitz C, Binder A, Groschel K, Hennerici MG, Lobotesis K, Poli S, Seidel G, Neumann-Haefelin T, Ringleb PA, Heuschmann PU, Veltkamp R. Safety of Endovascular Thrombectomy in Patients Receiving Non-Vitamin K Antagonist Oral Anticoagulants. Stroke. 2016 Apr;47(4):1127-30. doi: 10.1161/STROKEAHA.116.012684. Epub 2016 Mar 1. PMID 26931156
- See also: RASUNOA - Center Homepage — http://www.klinikum.uni-heidelberg.de/Schlaganfall-Studien.707.0.html